CLINICAL TRIAL: NCT05698459
Title: A Phase I, Open-label, Dose Escalation Study to Evaluate the Safety ,tolerance and Pharmacokinetics of OH2 Via Transcatheter Intraarterial Infusion in Patients with Advanced Liver Cancer
Brief Title: OH2 Oncolytic Viral Therapy Via Transcatheter Intraarterial Infusion in Patients with Advanced Liver Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH-OH2-011
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Advanced Liver Cancer
Keywords: Oncolytic Virus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OH2 (Experimental): Administration：intratumoral injection Frequency：once every 3 weeks
  Interventions: Biological: OH2 injection

INTERVENTIONS:
Biological: OH2 injection — OH2 injection administered by transcatheter Intraarterial infusion

SUMMARY:
An open-label dose-escalation phase I clinical study to evaluate the safety, tolerability and pharmacokinetics of OH2 injection via transcatheter Intraarterial infusion in patients with advanced hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood the study and voluntarily signed the informed consent (the informed consent must be signed before performing any procedure specified in the test);
2. Age 18-75 years old (inclusive);
3. Patients with primary or metastatic liver cancer confirmed histologically or cytologically;
4. Patients with liver cancer who have failed standard treatment, are not suitable for or are not willing to accept standard treatment;
5. ECOG physical condition 0 or 1;
6. Meet Child-Pugh liver function rating: Grade A or B;
7. Adequate bone marrow, liver, kidney and organ functions, meeting the following requirements in laboratory examination within 7 days prior to the first medication (no blood transfusion, blood products, no correction of granulocyte colony stimulating factor or other hematopoietic stimulating factors within 14 days prior to the laboratory examination) :

   * Neutrophil absolute count (ANC) ≥1.5×109/L, platelet ≥100×109/L, hemoglobin ≥90g/L;
   * Serum total bilirubin ≤3 times the upper limit of the normal reference range (3×ULN);
   * Alanine transaminase (ALT) and/or aspartate transaminase (AST) ≤5×ULN;
   * Serum creatinine ≤1.5×ULN or creatinine clearance ≥50mL/min (as calculated by Cockcroft-Gault formula);
   * International Normalized ratio (INR) ≤1.5 or partially activated prothrombin time (APTT) ≤1.5×ULN;
8. Subjects with chronic HBV infection must receive HBV-DNA < 500IU/ml and HBsAg positive patients must receive antiviral therapy according to the Guidelines for Chronic Hepatitis B Prevention and Treatment 2015 Edition. HCV-RNA positive patients must receive antiviral therapy according to the Hepatitis C Prevention and Treatment Guidelines 2015 Edition and have liver function within the normal range;
9. Recovery of AE associated with previous systemic chemotherapy, radical/extensive radiotherapy to National Cancer Institute General Adverse Event Term 5.0 (NCI CTCAE V5.0) ≤ Class 1 (except hair loss, non-clinically significant and asymptomatic laboratory abnormalities);
10. For subjects with herpes, 3 months after completion of herpes treatment;
11. Expected survival ≥12 weeks;
12. Fertile women must have a negative serum or urine pregnancy test within 7 days before the first dose. Fertile male or female patients volunteered to use effective contraceptive methods, such as dual screen contraception, condoms, oral or injectable contraceptives, and intrauterine devices, during the study period and within 90 days of the last study medication. All female patients will be considered fertile unless they have undergone natural menopause, artificial menopause or sterilization (e.g. hysterectomy, bilateral adnexectomy or irradiation of radioactive ovaries).
13. More than 4 weeks after the end of previous anti-tumor therapy (including endocrine, chemical/radiotherapy, targeted therapy) (more than 6 weeks after the treatment of nitrosourea and mitomycin chemotherapy);
14. Four weeks after major surgery;
15. At least one measurable or evaluable lesion was present according to RECIST1.1 criteria.

Exclusion Criteria:

1. A history of pleural effusion related to moderate or severe ascites, hemorrhagic esophageal varices, hepatic encephalopathy, or liver insufficiency within 6 months prior to screening;
2. Patients with large tumors - tumors >50% by liver volume and/or invading inferior vena cava;
3. Non-recovery to National Cancer Institute General Adverse Event Term 5.0 (NCI CTCAE V5.0) level 1 toxicity (excluding hair loss, non-clinically significant and asymptomatic laboratory abnormalities) due to prior antitumor therapy prior to initial administration of the study drug;
4. Other malignancies (except basal cell carcinoma or squamous cell carcinoma of the skin and carcinoma in situ of the cervix that have been effectively controlled) in the past 5 years;
5. For subjects with known central nervous system metastases, if they have received BMS in the past and their condition is stable (no evidence of imaging progression is seen at least 4 weeks before the first administration of the trial therapy, and any neurological symptoms have returned to baseline), repeated imaging examinations confirm no evidence of new BMS or the expansion of the original BMS. Participants who do not require steroid therapy at least 14 days before the initial administration of the trial therapy are eligible to participate in the trial. Subjects with cancerous meningitis should be excluded regardless of whether they are clinically stable;
6. Received standard anti-tumor therapy for liver cancer within 4 weeks before the first drug use, including surgery, interventional therapy, systemic therapy, radiotherapy and traditional Chinese medicine therapy (the instructions for traditional Chinese medicine therapy with clear anti-tumor indications, and a one-week washout period is enough before the first drug use);
7. Received radical radiotherapy (including more than 25% bone marrow radiotherapy) within 4 weeks prior to initial medication;
8. Have previously received similar drugs for antitumor therapy;
9. Received major surgical operations (the definitions of major surgical operations refer to Grade 3 and Grade 4 operations specified in the "Measures for the Clinical Application of Medical Technology" implemented on May 1, 2009) or unhealed wounds, ulcers and fractures within 4 weeks before the first drug use;
10. The subjects currently have active gastric and duodenal ulcers, ulcerative colitis and other digestive tract diseases, or active bleeding from unexcised tumors, or other conditions determined by the researchers that may cause digestive tract bleeding and perforation;
11. Patients with significant evidence or history of bleeding tendency within 2 months prior to initial medication (bleeding >30mL within 2 months, hematemesis, black feces, and hematochezia), hemoptysis (>5mL of fresh blood within 4 weeks), or thromboembolic events (including stroke events and/or transient ischemic attacks) within 12 months;
12. Cardiovascular disease of significant clinical significance, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within 6 months prior to initial medication; New York Heart Association (NYHA) Grade >2 for congestive heart failure; Left ventricular ejection fraction (LVEF) <50%; Primary cardiomyopathy, a history of clinically significant prolonged QTc interval, or QTc interval >470ms in women and >450ms in men during the screening period;
13. Severe and uncorrectable electrolyte abnormalities determined by the investigator to be clinically significant;
14. The patient had an active infection or developed an unexplained fever (body temperature >38.5oC) during screening and prior to initial administration;
15. Preparing for or having previously received allogeneic organ or bone marrow transplantation, including liver transplantation;
16. Subjects with a past or current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, or severe impairment of lung function that might interfere with the detection and management of suspected drug-related pulmonary toxicity;
17. Patients with active tuberculosis (TB) who are receiving anti-TB therapy or have received anti-TB therapy within 1 year prior to initial medication; Known human immunodeficiency virus (HIV) infection; The copy number of hepatitis B and hepatitis C virus was active.
18. Pregnant women (positive pregnancy test before medication) or breastfeeding women;
19. Known allergy to any herpes virus and OH2 inJ ingredients;
20. Any other medical condition, clinically significant metabolic abnormality (e.g., uncontrolled diabetes, thyroid dysfunction), physical abnormality, or laboratory abnormality, in which, in the investigator's judgment, there is reason to suspect that the patient has a medical condition or condition unsuitable for the study drug (e.g., the presence of epileptic seizures and the need for treatment), Or it could affect the interpretation of the findings, or put patients at high risk.
21. Received the corresponding experimental drugs in clinical trials of other unapproved or unmarketed drugs within 4 weeks before the first drug use;
22. As determined by the investigator, the subjects had other factors that might have led to the forced termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
DLTs (Dose Limiting Toxicity) | 3 weeks from the first administration
  Toxic reactions according to the NCI-CTCAE 5.0 grading standard that occur within 3 weeks from the first administration, are judged to be drug-related by the investigator, and meet the non-hematological toxicity and hematological toxicity conditions specified in the clinical protocol
MTD (Maximum Tolerance dose) | 2 years
  If ≥2/6 subjects developed DLT, the previous dose group was MTD

SECONDARY OUTCOMES:
Incidence of AE (Adverse Event) and SAE (Serious Adverse Event) | 2 years
  According to the NCI-CTCAE 5.0 grading standard
Objective Response Rate | 2 years
  The assessment result is the number and proportion of subjects with complete response + partial response.
Disease Control Rate | 2 years
  The assessment result is the number and proportion of subjects with complete response + partial response + stable disease.
OS (Overall Survival) | 2 years
  The overall survival for each patient receiving OH2 will be calculated.
PFS (Progression Free Survival) | 2 years
  Time after OH2 administration to clinical and radiographic disease progression will be evaluated.
Biodistribution and viral shedding | 2 years
  OH2 DNA copy
Immunogenicity | 2 years
  HSV-2 antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China